CLINICAL TRIAL: NCT04859465
Title: Albumin-bound Paclitaxel Combined With Liposomal Doxorubicin in the Treatment of Advanced or Unresectable Angiosarcoma--an Open, Single Arm, Multicenter Phase II Study
Brief Title: Albumin-bound Paclitaxel Combined With Liposomal Doxorubicin in the Treatment of Advanced or Unresectable Angiosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xing Zhang, Director of department of medical sarcoma and melanoma,Principal Investigator,Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Angiosarcoma
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Angiosarcoma Metastatic
MeSH Terms: interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abraxane combined with liposomal doxorubicin (Experimental): Abraxane combined with liposomal doxorubicin in the treatment of advanced or unresectable angiosarcoma
  Interventions: Drug: Abraxane combined with liposomal doxorubicin

INTERVENTIONS:
Drug: Abraxane combined with liposomal doxorubicin — Patients with advanced or unresectable angiogenic sarcoma who met the criteria of treatment failure received abraxane combined with liposomal doxorubicin regimen. Administration regimen: abraxane 220 mg / m2 D1 plus liposomal doxorubicin 35 mg / m2 D1, IV drip, 3 weeks as a cycle, until the disease progression or intolerable toxicity. Up to 8 cycles.

SUMMARY:
The purpose is to explore the efficacy and safety of the combination of albumin-bound paclitaxel and liposomal doxorubicin in the treatment of advanced or unresectable angiosarcoma.

DETAILED DESCRIPTION:
Soft tissue sarcoma (STS) is a relatively rare malignant tumor. In recent years, the disease has been increasing gradually. As an important biological feature of soft tissue sarcoma is local recurrence and distant metastasis, most patients die of distant metastasis. Despite the improvement of local control rate, more than 50% of patients died of unresectable or distant metastasis due to tumor progression. Doxorubicin and ifosfamide based chemotherapy is the standard first-line treatment for patients with relapsed / distant metastasis / unresectable advanced soft tissue sarcoma. For patients who fail or cannot tolerate first-line treatment, the choice of treatment is still limited. At present, some clinical patients who failed to receive standard treatment have tried to use the albumin-bound paclitaxel and liposomal doxorubicin regimen, with the ORR of 33% and PFS of about 8 months. As a new combination of chemotherapy drugs, more targeted phase II clinical studies are needed to evaluate the efficacy and safety of the new chemotherapy drugs in a variety of cancer species. In view of the above problems, this study aims to observe and explore the efficacy and safety of the combination of albumin-bound paclitaxel (keaili) and liposomal doxorubicin (duomeisu) in the treatment of advanced angiogenic sarcoma patients, and to provide better treatment options for patients with advanced sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. The patients voluntarily participated in the study and signed the informed consent; In all advanced angiogenic sarcomas confirmed by pathology, the standard treatment failed or there was no standard treatment or the standard treatment could not be tolerated. There is at least one measurable lesion according to RECIST 1.1, mainly including angiosarcoma, epithelioid hemangioendothelioma, epitheliosarcoma hemangioendothelioma, pseudomyogenic hemangioendothelioma, Kaposi sarcoma, malignant solitary fibroma / hemangiopericytoma, malignant glomus tumor, etc.
2. Patients in advanced stage with unresectable lesions or lymph node or distant metastasis by imaging evaluation;
3. In the past three months, there was at least one target lesion that could be measured according to RECIST version 1.1 standard, and it could be accurately measured in at least one direction (the maximum diameter needs to be recorded) by MRI or CT, including conventional CT ≥ 20 mm or spiral CT ≥ 10 mm.
4. 18-70 years old; ECOG PS score: 0-1; the expected survival time was more than 3 months;
5. The main organ function met the following criteria within 7 days before treatment (1) Blood routine examination standard (without blood transfusion within 14 days)

   * Hemoglobin (HB) ≥ 90g / L; ② Absolute neutrophil count (ANC) ≥ 1.5 × 109 / L;

     ③ Platelet count (PLT) ≥ 80 × 109 / L.

     (2) Biochemical tests should meet the following standards:
   * Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); ② Alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5 × ULN ALT and AST ≤ 5 ×ULN in patients with liver metastasis; ③ Serum creatinine (CR) ≤ 1.5 × ULN or creatinine clearance rate (CCR) ≥ 60ml / min;

     (3) Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ the lower limit of normal value (50%).
6. Women of childbearing age should agree to use contraceptive measures (such as intrauterine device, contraceptive or condom) during the study period and within 6 months after the end of the study; women with negative serum or urine pregnancy test within 7 days before the study and must be non lactation patients; men should agree to use contraceptive measures during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

1) Patients who have previously received abraxane treatment.

2) There were other malignant tumors in the past 5 years or at the same time, except for the cured cervical carcinoma in situ, skin cancer without melanoma and superficial bladder tumor (TA (non invasive tumor), tis (in situ cancer) and T1 (tumor infiltrating basement membrane);

3) Systemic anti-tumor treatment, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or mitomycin C use within 6 weeks prior to the treatment of the trial drug), is planned within 4 weeks before the group is given or during the study medication. The radiotherapy was performed within 4 weeks before the group or the limited field radiotherapy was performed within 2 weeks before the group;

4) With pleural effusion or ascites, respiratory syndrome (≥ CTC AE class 2 dyspnea (dyspnea 2 refers to shortness of breath when a small amount of activity is used; It can affect instrumental daily life activities);

5) No remission of toxic reactions caused by any previous treatment was higher than that of CTC AE (4.01), excluding hair loss and lymphocyte reduction;

6) Patients with any serious and / or uncontrollable diseases, including:

1. The patients with poor blood pressure control (systolic pressure ≥ 150 mmHg and diastolic pressure ≥ 100 mmHg) were found;
2. Patients with myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥ 480ms) and ≥ 2 congestive heart failure (NYHA classification);
3. Active or uncontrollable severe infection (≥ CTC AE Level 2 infection);
4. Cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis need to be treated with antiviral treatment;
5. Renal failure requires hemodialysis or peritoneal dialysis;
6. The control of diabetes mellitus was not good (FBG) was more than 10mmol/l;
7. The routine urine suggested that the urine protein was ≥ + +, and the 24-hour urine protein was more than 1.0 G;
8. Patients with epilepsy and need treatment;

7) The patients were treated with major surgery, incision biopsy or obvious traumatic injury within 28 days before entering the group;

8) Patients with any signs of bleeding constitution or history, regardless of severity; In the 4 weeks before entering the group, there were unconnected wounds, ulcers or fractures in patients with bleeding or bleeding events ≥ CTCAE Level 3;

9) The patients with arteriovenous thrombosis occurred within 6 months, such as cerebrovascular accidents (including transient ischemic attack), deep vein thrombosis and pulmonary embolism;

10) The patients with active ulcer, perforation and obstruction of intestine;

11) The patients had clinical symptoms of central nervous system metastasis (such as brain edema, hormone intervention, or brain metastasis progress); Patients who have received brain or meningeal metastasis treatment before, such as clinical stability (MRI) have been maintained for at least 2 months, and patients who have stopped systemic hormone therapy (dose > 10mg / day prednisone or other therapeutic hormone) for more than 2 weeks can be included;

12) The subjects were using immunosuppressant, or systemic or absorbable local hormone therapy to achieve immunosuppressive purposes (dose > 10mg / day prednisone or other therapeutic hormone), and were still in use within 2 weeks before entering the group;

13) The subjects had any active autoimmune disease or had a history of autoimmune disease (such as, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; If the subjects had vitiligo or had been completely relieved in childhood asthma, no intervention was needed in adult; Asthma in which the subjects needed bronchodilators to intervene in medicine could not be included;

14) Subjects had active tuberculosis and immunodeficiency history including human immunodeficiency virus (HIV) or other acquired or congenital immunodeficiency disease or active hepatitis (transaminase does not conform to inclusion, hepatitis B virus (HBV) DNA ≥ 104/ ml or hepatitis C virus seropositive (HCV) RNA ≥ 103/ml or higher); Chronic hepatitis B virus carriers with HBV DNA < 2000 iu/ml (< 104 / ml) must be treated with antiviral therapy throughout the study.

15) According to the researchers' judgment, the subjects are not suitable for entering the group or other factors may lead to the termination in the middle of the course. For example, other serious diseases (including mental diseases) need to be treated together, there are serious laboratory abnormalities, and family or social factors, which will affect the safety of the subjects, or the collection of test data and samples;

16) The clinical trials of other anti-tumor drugs were conducted 28 days before entering the group.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 24 months
  Overall response rate (ORR) of patients with advanced or unresectable angiosarcoma treated with abraxane combined with liposomal doxorubicin

CONTACTS AND LOCATIONS:
Overall Officials: Xing Zhang, Principal Investigator — Sun Yat-sen University CancerCenter
Locations (1):
- Xing Zhang, Guangzhou, Guangdong, China